CLINICAL TRIAL: NCT05600140
Title: Viewing Strategy Training in Children With (Cerebral) Visual Impairment: From Spontaneous Eye Movements to a Structured Viewing Strategy
Brief Title: Viewing Strategy Training in Children With (Cerebral) Visual Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Dutch Visio (Other)
Collaborators: Radboud University, Behavioural Science Institute, Nijmegen, The Netherlands (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81584.091.22
Record Dates: First submitted 2022-07-12; First posted 2022-10-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Vision Disorders; Vision, Low
Keywords: viewing strategies; (cerebral) visual impairment; visual rehabilitation; reading strategies; visual search strategies
MeSH Terms: conditions — Vision Disorders; Vision, Low; Blindness, Cortical

STUDY DESIGN:
Intervention Model Description: For the first phase of the study, we aim to include 48 children aged 5-12 years for each group (i.e. normal Vision, ocular visual impairment, cerebral visual impairment). For the second phase of the study 60 children with visual impairment aged 5-9 years will be included (ocular impairment: n=30, cerebral visual impairment: n=30).
  In the second phase of the project, children receive a visual training of viewing strategies (six weeks, 2 times a week, 30 minutes). During the training, children are instructed to use specific viewing strategies (looking in a structured direction which fits the task at hand, zooming in and out / change of visual selective attentional field, visual discrimination). The verbal instructions and exercises are protocol based. A textbook is used to describe the reactions of the children during training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A) early training group (Experimental): T0 = baseline measurement T1 = posttest (within two weeks after training) T2 = follow up measurement (6 months after training)
  Interventions: Behavioral: Viewing strategy training
- Group B) late training group (Experimental): T0 = baseline measurement T1 = test-retest reliability and natural development (over period 1 1/2-2 months after T0) T2 = posttest (within two weeks after training)
  Interventions: Behavioral: Viewing strategy training

INTERVENTIONS:
Behavioral: Viewing strategy training — Children receive a visual training of viewing strategies (six weeks, 2 times a week, 30 minutes). During the training, children are instructed to use specific viewing strategies (looking in a structured direction which fits the task at hand, zooming in and out / change of visual selective attentional field, visual discrimination). The verbal instructions and exercises are protocol-based. A textbook is used to describe the reactions of the children during training.

SUMMARY:
Viewing strategies are strategies used to process visual Information. Many children with visual impairment seem to lack systematic viewing strategies. However, it is unknown how viewing strategies differ between children with normal vision and children with (cerebral) visual impairment. In addition, viewing strategy training is often adopted in clinical practice, but till date there is no scientific evidence about effectiveness of this approach.

The current project has two goals: (1) to measure viewing strategies used by children with normal vision, children with ocular visual impairment and children with CVI, and (2) to evaluate whether training viewing strategies results in more efficiënt visual Information processing.

ELIGIBILITY:
Inclusion criteria typically developing children with normal vision:

* Age 5-12 years
* linear distant visual acuity of 0.1 logMAR or better
* Verbal IQ above 70
* Absence of developmental disorders or psychiatric problems like ASS or AD(H)D

Inclusion criteria for children with ocular visual impairment:

* Age 5-12 years
* Children with linear distance visual acuity better <=1.3logMAR and >0.1 logMAR
* Intact central visual field (at least > 30 degrees)
* Children with a verbal IQ above 70
* Absence of developmental disorders or psychiatric problems like ASS or AD(H)D

Inclusion criteria for children with cerebral visual impairment:

* Age 5-12 years
* Linear distance visual acuity <=0.3 logMAR
* Having the diagnosis CVI (verified by ophthalmologists)
* Children with a verbal IQ above 70
* Absence of psychiatric problems like ASS or AD(H)D

Additional inclusion criterion for study 2 (evaluating training effectiveness): children with (cerebral) visual impairment should have an indication for viewing strategy training. Training should not be indicated if children have no problems performing academic tasks (i.e. when speed and accuracy of visual processing is within the normal range). The age range for study 2 is 5-9 years.

Exclusion criteria:

* Children with VI: linear near visual acuity >1.0 logMAR
* Children with visual field defect < 30 degrees
* Children with a verbal IQ below 70
* Children who attended a form of vision training in the past two years
* Children with psychiatric problems like ASS or AD(H)D
* Auditory impairment or language impairments
* Major life events during training

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in reading accuracy after viewing strategy training | Group A: Day 0, Month 2, Month 8; group B: Day 0, Month 2, Month 4
  Radner reading test
Changes in reading speed after viewing strategy training | Group A: Day 0, Month 2, Month 8; group B: Day 0, Month 2, Month 4
  Radner reading test
Changes in visual search accuracy after training | Group A: Day 0, Month 2, Month 8; group B: Day 0, Month 2, Month 4
  Accuracy during conjunction search
Changes in visual search speed after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  Speed during conjunction search
Changes in saccade amplitudes during reading and visual search after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  Saccade amplitudes measured using Radner reading test and conjunction search
Changes in fixation duration during reading and search after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  Fixation durations measured using Radner reading test and conjunction search
Changes in average distance between fixation points during conjunction search (EB-VSA) after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  Average distance between fixation points using Radner reading test and conjunction search

SECONDARY OUTCOMES:
Changes in WISC-V visual processing speed index (VSI) after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  WISC-IV visual processing speed index
Changes in local visual selective attention after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  TEA-Ch Speurtocht (total number of symbols found in 1 minute)
Changes in global visual selective attention after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  Gestalt Closure (Kaufman-ABC), number of correct answers
Changes in visual identification speed after training | Group A: Day 0, Month 2, Month 8; Group B: Day 0, Month 2, Month 4
  'DST-Plaatjes Benoemen', number of pictures correctly named within 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Huurneman, PhD, Principal Investigator — Royal Dutch Visio
Locations (1):
- Royal Dutch Visio, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No